CLINICAL TRIAL: NCT02535637
Title: Impact of Breastfeeding and Obesity on Offspring Body Composition and Growth at Six Months of Age
Brief Title: Breastfeeding and Obesity on Offspring Body Composition
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Collaborators: Mead Johnson Nutrition (Industry)
Responsible Party: Principal Investigator, David A. Fields, PhD, Associate Professor, University of Oklahoma
Other Study IDs: 15246
Record Dates: First submitted 2015-08-24; First posted 2015-08-28 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Obesity; Breast Milk Collection
MeSH Terms: conditions — Obesity; Breast Milk Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mothers-Infant: Mothers who were planning to exclusively breastfeed for six months were enrolled into the study along with their infant.
  Interventions: Other: Exclusively breastfeed

INTERVENTIONS:
Other: Exclusively breastfeed — There is no intervention other than mothers must exclusively breastfeed.

SUMMARY:
The purpose of this study is to explore the effect maternal obesity and breastfeeding play on infant body composition. The investigators hypothesize in the first 6 months of life breast fed offspring from overweight / obese mothers will be fatter with greater trunk fat mass and accumulate fat at a greater rate than breast fed infants from normal weight mothers. Furthermore, the investigators postulate that circulating maternal milk adipocytokines will positively correlate to total fat mass at six months of age.

DETAILED DESCRIPTION:
The objective of this study is to determine if offspring from overweight/obese non-diabetic mothers whom breastfeed have greater total fat and trunk fat mass and accumulate fat mass at a greater rate from ~ 1 month to 6 months of life compared to breastfed infants from normal weight mothers.

Specific Aim 1: Understand how maternal obesity and breast-feeding impact body composition of the offspring. Based upon the investigators preliminary data and counter to accepted dogma the hypothesis is at six months of age total fat mass, particularly in the trunk will be elevated at 6 months of age in infants whose mother was either overweight or obese vs. infants from normal weight mothers.

Specific Aim 2: Identify adipocytokines in breast milk. The postulate is breast milk from overweight and obese mothers will have greater levels of insulin, glucose, Ghrelin, IGF-1, IL-6, TNFα, high-sensitivity C-reactive protein, and lower Leptin levels than breast milk from normal weight mothers and will be correlated with offspring fat mass.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 37 and 41 weeks
* Singleton birth
* Infant in good health
* 40±5 days old at enrollment
* Infant is being exclusively breastfed (defined as fed directly from the breast or with mother's expressed milk and receiving no formula in the last 20 days prior to enrollment)
* Mother of an infant being exclusively breastfed plans to continue this exclusive feeding from the time of enrollment until six months of age
* Parent/caregiver demonstrates an understanding of the given information and ability to record the requested data
* Having obtained informed consent of legal representative

Exclusion Criteria:

* Congenital illness or malformation that affects infant feeding and/or growth
* Significant pre-natal and/or post-natal disease
* Infant has received any complementary feeding, i.e. any nutrition besides breast milk
* In the investigators assessment, infant's family cannot be expected to comply with treatment (feeding regimen)
* Currently participating in another clinical trial

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 37 mothers whom exclusively breast fed to six-months. Participants (mothers/infant) included offspring from mothers with a singleton-term healthy pregnancy (37-40 weeks). Both vaginal and cesarean deliveries were included. Infants who are exclusively breastfed (defined as no formula in the last 20 days) prior to enrollment will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2010-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The association of breast milk adipocytokines with maternal body mass index at one and 6-months of age. | One to 6-months.
  The associations between breast milk adipocytokines and maternal fatness (i.e. body mass index) will be determined at both one and 6-months.
The association of breast milk adipocytokines with infant body composition at one and 6-months of age. | One to 6-months.
  The associations between breast milk adipocytokines and infant body composition (i.e. total fat and fat-free mass and the percentage of body fat) will be determined at both one and 6-months.

SECONDARY OUTCOMES:
The change in infant body composition (body fat and fat-free mass) from one to 6-months of age. | One to 6-months.
  The change in infant body composition will be measured from 1 to 6-months. Body composition is defined as the change (in grams) in total fat mass, total fat-free mass and the percentage of fat mass (%fat).
The change in breast milk adipocytokines levels from one to 6-months. | One to 6-months.
  The change in leptin (pg/mL), insulin (pg/mL), glucose (mg/mL), ghrelin (pg/mL), IGF-1 (pg/mL), IL-6 (pg/mL), TNFα (pg/mL), high-sensitivity C-reactive protein (pg/mL) will be determined in breast milk from one and 6-months.

CONTACTS AND LOCATIONS:
Overall Officials: David A Fields, PhD, Principal Investigator — Faculty

REFERENCES:
- [Derived] Wolfs D, Lynes MD, Tseng YH, Pierce S, Bussberg V, Darkwah A, Tolstikov V, Narain NR, Rudolph MC, Kiebish MA, Demerath EW, Fields DA, Isganaitis E. Brown Fat-Activating Lipokine 12,13-diHOME in Human Milk Is Associated With Infant Adiposity. J Clin Endocrinol Metab. 2021 Jan 23;106(2):e943-e956. doi: 10.1210/clinem/dgaa799. PMID 33135728
- [Derived] Isganaitis E, Venditti S, Matthews TJ, Lerin C, Demerath EW, Fields DA. Maternal obesity and the human milk metabolome: associations with infant body composition and postnatal weight gain. Am J Clin Nutr. 2019 Jul 1;110(1):111-120. doi: 10.1093/ajcn/nqy334. PMID 30968129
- [Derived] Fields DA, George B, Williams M, Whitaker K, Allison DB, Teague A, Demerath EW. Associations between human breast milk hormones and adipocytokines and infant growth and body composition in the first 6 months of life. Pediatr Obes. 2017 Aug;12 Suppl 1(Suppl 1):78-85. doi: 10.1111/ijpo.12182. Epub 2017 Feb 3. PMID 28160457
- [Derived] Alderete TL, Autran C, Brekke BE, Knight R, Bode L, Goran MI, Fields DA. Associations between human milk oligosaccharides and infant body composition in the first 6 mo of life. Am J Clin Nutr. 2015 Dec;102(6):1381-8. doi: 10.3945/ajcn.115.115451. Epub 2015 Oct 28. PMID 26511224